CLINICAL TRIAL: NCT03937531
Title: Comparison of Postoperative Voiding Dysfunction in Two Voiding Trials After Retropubic Midurethral Slings: a Randomized Controlled Trial
Brief Title: Void Trials After Two Voiding Trials (TVT)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI Left the Institution
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Woojin Chong-Kaufman, Assistant Professor & Assistant FPMRS Program Director, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GCO 19-0816
Record Dates: First submitted 2019-05-02; First posted 2019-05-03 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Postoperative Voiding Dysfunction; Postoperative Urinary Retention
Keywords: Postoperative voiding dysfunction; Postoperative void trial; Retrograde fill void trial; Spontaneous void trial; Midurethral sling

STUDY DESIGN:
Intervention Model Description: Subjects will be enrolled consecutively during either the surgical preoperative evaluation or in the preoperative holding area before surgery. Participation in the study would not alter their surgical treatment plan. Randomization will be determined through computer-generated random number blocks of six. A sequentially numbered, opaque, sealed envelope will be opened for each subject after the recruitment and consenting process, and subjects will be assigned to one of two groups: retrograde fill void trial (RVT) vs spontaneous void trial (SVT).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retrograde-fill void trial (RVT) (Experimental): Subjects will leave the operating room with a urinary catheter inserted. Subjects should be recovered from anesthesia effects (2-3 hours after surgery) before voiding trial. First, the bladder will be completely drained into the Foley bag then the bag will be detached from the catheter. The bladder will be back-filled with sterile water (300 mL). After the catheter is removed, subjects are expected to void at least 2/3 (200 mL) of the total instilled amount within 30 minutes of filling. Post-void residual (PVR) will be measured by both subtraction of the voided volume from 300cc and by using a bladder scanner.
  Interventions: Procedure: Bladder Scanner
- Spontaneous void trial (SVT) (Active Comparator): Subjects will leave the operating room without a urinary catheter. Participants are allowed up to 6 hours after surgery for spontaneous voiding. After voiding, the voided volume will be noted. PVR will be measured using a bladder scanner.
  In both groups, if PVR >=100 mL on a bladder scanner, an indwelling urinary catheter will be placed and the actual PVR will be documented. Subjects who failed voiding trial will be instructed to return to clinic within 2-4 days for the second void trial. Prophylactic antibiotics will NOT be given. The time to discharge will be measured for each subject. This will be determined by calculating the time between arrival to the PACU and the time of discharge using documentation from EPIC.
  Interventions: Procedure: Bladder Scanner

INTERVENTIONS:
Procedure: Bladder Scanner — PVR will be measured by using a bladder scanner.

SUMMARY:
The primary objective of this project is to compare the rate of postoperative voiding dysfunction in two voiding trials (the retrograde-fill technique versus the spontaneous-fill technique) after midurethral sling (MUS) procedures with tension-free vaginal tape (TVT) without any concomitant surgery.

DETAILED DESCRIPTION:
The purpose of this research study is that the study investigators want to find out if there is a way of reducing patients' postoperative emotional stress from having a separate procedure to test their urinary function after "sling" surgery. Women with stress urinary incontinence (leakage of urine with physical activities like coughing, jumping, running, laughing, etc) may need "sling" surgery to help their urinary leakage problems. "Sling" surgeries in our hospital are mainly done using a retropubic midurethral sling (sling is passed to the space in front of your bladder). It is well known that having a sling surgery dramatically helps women with stress urinary incontinence. However, any surgical managements can have complications. One of the common complications from having a sling is "postoperative voiding dysfunction". In other words, some women may have a problem with urinating normally after the sling surgery. The most common problem is that some women (up to 4 out of 10 women) may not be able to urinate right after the surgery for the brief period of the time. The study team calls this condition "urinary retention". Postoperative urinary retention after the sling surgery can occur mainly due to pain, anesthesia effect, underlying tissue swelling; and rarely secondary to bleeding or nerve damage. Not being able to urinate for long time (>6-8 hours) can damage the bladder muscle and nerves to the bladder. Therefore, most surgeons like to perform a "bladder testing" in the recovery unit before you are ready to go home to make sure you would be able to urinate at home once discharged. Traditionally, the bladder testing is involved with back-filling the bladder with sterile water (about 300cc) and checking if the patients are able to urinate within 30 minutes. The patients should be able to urinate about two thirds of amount that has been placed in the bladder. This "bladder testing" can create a lot of emotional stress to the patients; consequently, some of the patients may not be able to urinate within the given time although there is nothing wrong with their bladder function. Those patients, who did not pass this testing, are sent home with an indwelling urinary catheter with legbag until they come back to clinic for another "bladder testing" in 3-7 days. It is well known that the indwelling catheters are a leading cause of urinary tract infection and a source of patients' discomfort, embarrassment, and inconvenience. Therefore, this study is designed to find out if having a bladder test after the sling surgery is a really-must thing to perform to test the bladder function. The study team would like to investigate if allowing the patients to have enough time to urinate their own, without making them to go through the bladder testing, would be a sufficient way of testing the bladder function after sling surgery.

ELIGIBILITY:
Inclusion Criteria:

* Any adult female (age >= 18 years old) undergoing an outpatient TVT surgery for SUI will be eligible for participation.
* Participants must be able to provide informed consent and complete all study requirements.

Exclusion Criteria:

* Participants will be excluded if the surgery involves any concomitant urinary tract or pelvic reconstructive procedure or if the procedure, in itself, necessitates PUC, as in the event of a cystotomy, bladder perforation or intraoperative hemorrhage
* Participants with a history of neurologic conditions affecting the urinary tract system, POP beyond the hymen during straining (any compartment), or previous anti-incontinence procedure will be also excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2020-02 (Estimated); Primary Completion 2021-05-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Void trial failure rates | Day of surgery
  The void trial failure rates requiring postoperative urinary catheterization after midurethral sling procedures with transvaginal tape (TVT) without concomitant surgery. First, the bladder will be completely drained into the Foley bag then the bag will be detached from the catheter. The bladder will be back-filled with sterile water (300 mL).
  After the catheter is removed, subjects are expected to void at least 2/3 (200 mL) of the total instilled amount within 30 minutes of filling. PVR will be measured by both subtraction of the voided volume from 300cc and by using a bladder scanner.

SECONDARY OUTCOMES:
Number of participants with Postoperative urinary retention (POUR) | 2 weeks and 6 weeks post surgery
  POUR any time up to 6 weeks after surgery: after discharge, subjects will be monitored for any encounters for POUR and will be asked at 2 weeks and 6 weeks post-operative visit if they have had a catheter placed outside the hospital. Additionally, any subject who fails their 2nd void trial will be noted.
Time to discharge | On the day of surgery
  Time to discharge will be determined by calculating the time between arrival to the PACU and the time of discharge using documentation from EPIC. Time to discharge is expected to happen on the day of surgery regardless of success or failure of void trial.
Number of participants with Urinary tract infection | Within 6 weeks after surgery
  UTI any time up to 6 weeks after surgery: subjects with a culture-proven UTI or >= 2 urinary symptoms (urinary urgency, frequency, dysuria, suprapubic pain, foul-smelling urine) plus pyuria on urine dip or urine analysis will be noted. Antibiotic treatment will be noted.
Incontinence Severity Index (ISI) | 2 weeks and 6 weeks post surgery
  ISI total scored from 0-12, with higher score indicating more severity of symptoms.
Urogenital Distress Inventory short form (UDI-6) | 2 weeks and 6 weeks post surgery
  UDI-6 is a 6 -item questionnaire, each item scored 0-3 with total score from 0 to 0 to 75, with higher score indicating more distress.
Patient Global Impression of Improvement (PGI-I) | 2 weeks and 6 weeks post surgery
  PGI-I is scored on a 7 likert score, with total score from 1 to 7, with higher score indicating worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Woojin Chong, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Mount Sinai West, New York, New York
  - Mount Sinai Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosseland LA, Stubhaug A, Breivik H. Detecting postoperative urinary retention with an ultrasound scanner. Acta Anaesthesiol Scand. 2002 Mar;46(3):279-82. doi: 10.1034/j.1399-6576.2002.t01-1-460309.x. PMID 11939918
- [Background] Partoll LM. Efficacy of tension-free vaginal tape with other pelvic reconstructive surgery. Am J Obstet Gynecol. 2002 Jun;186(6):1292-5; discussion 1295-8. doi: 10.1067/mob.2002.123736. PMID 12066111
- [Background] Tunitsky-Bitton E, Murphy A, Barber MD, Goldman HB, Vasavada S, Jelovsek JE. Assessment of voiding after sling: a randomized trial of 2 methods of postoperative catheter management after midurethral sling surgery for stress urinary incontinence in women. Am J Obstet Gynecol. 2015 May;212(5):597.e1-9. doi: 10.1016/j.ajog.2014.11.033. Epub 2014 Nov 27. PMID 25434837
- [Background] Trautner BW, Darouiche RO. Catheter-associated infections: pathogenesis affects prevention. Arch Intern Med. 2004 Apr 26;164(8):842-50. doi: 10.1001/archinte.164.8.842. PMID 15111369
- [Background] Barron KI, Savageau JA, Young SB, Labin LC, Morse AN. Prediction of successful voiding immediately after outpatient mid-urethral sling. Int Urogynecol J Pelvic Floor Dysfunct. 2006 Nov;17(6):570-5. doi: 10.1007/s00192-005-0064-8. Epub 2006 Apr 1. PMID 16583182
- [Background] Geller EJ. Prevention and management of postoperative urinary retention after urogynecologic surgery. Int J Womens Health. 2014 Aug 28;6:829-38. doi: 10.2147/IJWH.S55383. eCollection 2014. PMID 25210477
- [Background] Luber KM. The definition, prevalence, and risk factors for stress urinary incontinence. Rev Urol. 2004;6 Suppl 3(Suppl 3):S3-9. PMID 16985863
- [Background] Barber MD, Kleeman S, Karram MM, Paraiso MF, Walters MD, Vasavada S, Ellerkmann M. Transobturator tape compared with tension-free vaginal tape for the treatment of stress urinary incontinence: a randomized controlled trial. Obstet Gynecol. 2008 Mar;111(3):611-21. doi: 10.1097/AOG.0b013e318162f22e. PMID 18310363
- [Background] Dieter AA, Amundsen CL, Visco AG, Siddiqui NY. Treatment for urinary tract infection after midurethral sling: a retrospective study comparing patients who receive short-term postoperative catheterization and patients who pass a void trial on the day of surgery. Female Pelvic Med Reconstr Surg. 2012 May-Jun;18(3):175-8. doi: 10.1097/SPV.0b013e3182544e03. PMID 22543772
- [Background] Yokoe DS, Anderson DJ, Berenholtz SM, Calfee DP, Dubberke ER, Ellingson KD, Gerding DN, Haas JP, Kaye KS, Klompas M, Lo E, Marschall J, Mermel LA, Nicolle LE, Salgado CD, Bryant K, Classen D, Crist K, Deloney VM, Fishman NO, Foster N, Goldmann DA, Humphreys E, Jernigan JA, Padberg J, Perl TM, Podgorny K, Septimus EJ, VanAmringe M, Weaver T, Weinstein RA, Wise R, Maragakis LL; Society for Healthcare Epidemiology of America (SHEA). A compendium of strategies to prevent healthcare-associated infections in acute care hospitals: 2014 updates. Infect Control Hosp Epidemiol. 2014 Aug;35(8):967-77. doi: 10.1086/677216. PMID 25026611
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- See also: Oliphant SS, Wang L, Bunker CH, Lowder JL. Trends in stress urinary incontinence inpatient procedures in the United States, 1979-2004. Am J Obstet Gynecol. 2009; 200: 521.e1-521.e6 — http://dx.doi.org/10.1016/j.ajog.2009.01.007
- See also: EL-Hefnawy A, Wadie B, Abed A, Nabeeh A. Post-operative complications of midurethral slings: is it possible to use Clavien's classification? [ICS Abstract 848]. — https://www.ics.org/Abstracts/Publish/106/000848.pdf
- See also: Elkadry EA, Kenton KS, FitzGerald MP, Shott S, Brubaker L. Patient-selected goals: a new perspective on surgical outcome. Am J Obstet Gynecol. 2003; 189: 1551-1558. — https://doi.org/10.1016/S0002-9378(03)00932-3